CLINICAL TRIAL: NCT01640210
Title: TECHNICAL EVALUATION OF JEWELPUMP IN TYPE 1 DIABETIC PATIENTS TREATED WITH EXTERN INSULIN PUMP
Acronym: DIABELOOP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre d'Etudes et de Recherche pour l'Intensification du Traitement du Diabète (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2011-A00666-35
Record Dates: First submitted 2012-06-25; First posted 2012-07-13 (Estimated); Last update posted 2012-07-13 (Estimated); Status verified 2011-12

CONDITIONS: Type1diabetes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: JewelPUMP (insulin patch pump) — The study will be proposed during the visit of selection.
  Visit of inclusion:
  This visit will take place after having received the consent of the patient. Women will be asked to achieve a pregnancy test. Patients will wear a JewelPUMP containing saline solution in parallel with their usual insulin pump. They will be trained to use JewelPUMP.
  Patients treated with insulin pump will be instructed to reproduce the same "programming" between their usual pump and the JewelPUMP, they will use in parallel.
  Volume infused will be evaluated during a period of basal and bolus with a precision scale.
  Patient monitoring: Patient have to come back to the centre every 24 hours for 3 days. Study visit:
  Patients will be asked to fill out a questionnaire of satisfaction to the JewelPUMPTM and Visual scales.
  Volume infused will be evaluated with a precision scale, by comparison of weight of JewelPUMP and patients' usual pump

SUMMARY:
The main objective of the study is to verify the reliability of the solutes volumes issued by the Debiotech JewelPUMPTM controlled by its remote.

Three clinical sites are participating in this study:

* CHSF, Service of Endocrinology and Diabetology, CORBEIL-ESSONNES (91): Dr. Guillaume CHARPENTIER, Dr. Sylvia FRANC
* Grenoble University Hospital, Department of Endocrinology, Diabetes Diseases, Nutrition, GRENOBLE (38): Pr Pierre-Yves BENHAMOU
* CHU Jean Minjoz, Department of Endocrinology and Diabetology, BESANCON (25): Professor Alfred PENFORNIS, Dr. Annie CLERGEOT

The study will be conducted in 20 patients with type 1 diabetes treated by external insulin pump. Patients will be informed of the study during a screening visit. After signing the informed consent, they will return to the center where they will wear a JewelPUMPTM containing saline water, they will use their pumps in parallel. The investigator or nurse education will form the operation of the JewelPUMPTM and they will be instructed to replicate the same settings between their usual and JewelPUMPTM pump. The patient will be asked to complete visual analog scales of satisfaction with their usual treatment and the various elements of the devices (usual pump, and JewelPUMPTM) have been weighed using a precision balance to have a form of a base for comparison.

Patients will leave home for a period of about three days, but they will have to come back every days to the center. They will be asked to collect all events arising (programming problems to deliver a bolus, hardware failure ...) in a booklet.

At the end of study visit, patients will return to the center where the volumes will be assessed by the perfused weighed the various components and devices where they will complete the visual analog scales of satisfaction at endpoint.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 Diabetic patient treated by external insulin pump for at least 6 months
* Patient with a HbA1c < 9%
* Patient age over 18 years of age
* Patient having signed the consent and informed form
* Patient affiliated with the social security

Exclusion Criteria:

* Patients with diabetes type 2
* Patient pregnant or likely to be
* All serious pathologies that can interfere with the study
* Incompatible psychiatric pathologies with the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2011-11; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
weight of the insulin pump (JewelPUMP and usual pump) | 3 Days
  accuracy of volume delivered by the JewelPUMP by comparison of the difference of weight between usual pump and JewelPUMP at Day 1, Day 2 and day 3.

SECONDARY OUTCOMES:
satisfaction of patients | 3 days
  the satisfaction of the JewelPUMP for the patients is evaluated with visual analogic scales.
  patients indicate the their satisfaction of the JewelPUMP on a scale of 10 centimeter. on the left = no satisfaction and on the right = 100% satisfaction.
handling | 3 days
  the workability of the JewelPUMP for the patients is evaluated with visual analogic scales.
  patients indicate the workability of the JewelPUMP on a scale of 10 centimeter. on the left = no workability and on the right = 100% workability.
acceptability | 3 days
  the acceptability of the JewelPUMP for the patients is evaluated with visual analogic scales.
  patients indicate the acceptability of the JewelPUMP on a scale of 10 centimeter. on the left = no acceptability and on the right = 100% acceptability.

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume Charpentier, MD, Principal Investigator — CHSF
Locations (2):
- France (2):
  - CHU Jean Minjoz, Besançon
  - University Hospital Grenoble, Grenoble